CLINICAL TRIAL: NCT01628393
Title: A Phase 2/3, Multi-center, Randomized, Double-blind, Placebo-controlled (Part A) and Double-blind, Double-dummy, Active-controlled (Part B), Parallel Group Study to Evaluate the Efficacy and Safety of RPC1063 Administered Orally to Relapsing Multiple Sclerosis Patients
Brief Title: Efficacy and Safety Study of Ozanimod (RPC1063) in Relapsing Multiple Sclerosis Patients
Acronym: RADIANCE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RPC01-201-PartA; 2012-002714-40 (EudraCT Number)
Record Dates: First submitted 2012-06-22; First posted 2012-06-26 (Estimated); Results first posted 2021-02-11 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-01

CONDITIONS: Relapsing Multiple Sclerosis
MeSH Terms: interventions — ozanimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ozanimod 0.5 mg (Experimental): Participants received ozanimod 0.5 mg oral capsules daily for 24 weeks. Participants who completed the 24-week treatment period had the option to enter the blinded extension period and continue to receive ozanimod 0.5 mg weekly for another 96 weeks.
  Interventions: Drug: Ozanimod
- Ozanimod 1 mg (Experimental): Participants received ozanimod 0.5 mg oral capsules daily for 24 weeks. Participants who completed the 24-week treatment period had the option to enter the blinded extension period and continue to receive ozanimod 1 mg weekly for another 96 weeks.
  Interventions: Drug: Ozanimod
- Placebo (Placebo Comparator): Participants received placebo to ozanimod oral capsules daily for 24 weeks. Participants who completed the 24-week treatment period had the option to enter the blinded extension period and were randomized to receive ozanimod 0.5 mg or 1 mg weekly for 96 weeks.
  Interventions: Drug: Ozanimod; Drug: Placebo

INTERVENTIONS:
Drug: Ozanimod — Oral capsule taken once a day
  Other Names: RPC1063; Zeposia®
Drug: Placebo — Oral capsule taken once a day
  Arms: Placebo

SUMMARY:
This study is a two-part trial consisting of Part A (presented in this record) and Part B (see NCT02047734).

The primary objective in Part A of this study was to demonstrate the superior efficacy of ozanimod compared to placebo by showing a reduction in the cumulative number of total gadolinium-enhancing (GdE) lesions from Week 12 to Week 24 in patients with relapsing multiple sclerosis (RMS).

ELIGIBILITY:
Inclusion Criteria:

* Multiple sclerosis as diagnosed by the revised 2010 McDonald criteria
* Expanded Disability Status Scale (EDSS) score between 0 and 5.0 at Baseline

Exclusion Criteria:

* Secondary or primary progressive multiple sclerosis

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 258 (Actual)
Dates: Start 2012-09-18 (Actual); Primary Completion 2014-04-13 (Actual); Study Completion 2016-05-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (58):
- United States (6):
  - Alta Bates Summit Medical Center, Berkeley, California
  - Neuro Pain Medical Center, Fresno, California
  - University of California Davis Medical Center, Sacramento, California
  - The Neurological Institute PA, Charlotte, North Carolina
  - Neurology and Neuroscience Associates Inc., Akron, Ohio
  - The Polyclinic, Seattle, Washington
- Belgium (3):
  - Cliniques Universitaires St-Luc, Brussels
  - Centre Hospitalier Chretien Clinique Saint Joseph, Montegnée
  - Clinique Saint-Pierre, Ottignies
- University Multiprofile Hospital for Active Treatment Sv Ivan Rilski EAD, Sofia, Bulgaria
- Georgia (3):
  - Sarajishvili Institute of Neurology, Tbilisi
  - LTD MediClubGeorgia, Tbilisi
  - Khechinashvili University Hospital, Tbilisi
- Greece (3):
  - Evaggelismos General Hospital, Athens
  - 401 Military Hospital of Athens, Athens
  - Georgios Papanikolaou General Hospital of Thessaloniki, Thessaloniki
- Vaszary Kolos Korhaz, Esztergom, Hungary
- Azienda Ospedaliero Universitaria Policlinico Vittorio Emanuele, Cantania, Italy
- Poland (19):
  - Powiatowy Zespol Zakladow Opieki Zdrowotnej Szpital w Czeladzi, Czeladź
  - Regionalny Szpital Specjalistyczny im. dr Wladyslawa Bieganskiego, Grudziądz
  - Novo-Med Zielinski i wsp. Sp.J., Katowice
  - NEURO- CARE Site Management Organization Gabriela Klodowska-Duda, Katowice
  - NEURO MEDIC Janusz Zbrojkiewicz, Katowice
  - RESMEDICA Spolka z o.o., Kielce
  - Centrum Kompleksowej Rehabilitacji Sp.z.o.o. Szpital Wielospecjalistyczny, Konstancin-Jeziorna
  - Centrum Neurologii Krzysztof Selmaj, Lódzkie
  - Prof. dr med. Zbigniew Stelmasiak Specjalistyczny Gabinet Neurologiczny, Lublin
  - Wojewodzki Szpital Specjalistyczny, Olsztyn
  - Neurologiczny NZOZ Centrum Leczenia SM Osrodek Badan Klinicznych Dr n med Hanka Hertmanowska, Plewiska
  - Niepubliczny Zaklad Opieki Zdrowotnej KENDRON, Podlaskie
  - Niepubliczny Zaklad Opieki Zdrowotnej NEUROKARD Ilkowski i Partnerzy Spolka Partnerska Lekarzy, Poznan
  - EUROMEDIS Sp. z.o.o., Szczecin
  - Indywidualna Specjalistyczna Praktyka Lekarska Zbigniew Cebulski, Warminsko-mazurskie
  - Szpital Czerniakowski Samodzielny Publiczny Zaklad Opieki Zdrowotnej, Warsaw
  - Wojskowy Instytut Medyczny, Warsaw
  - Centralny Szpital Kliniczny MSWIA, Warsaw
  - Instytut Psychiatrii i Neurologii, Warsaw
- Romania (4):
  - Health Club Medical Center S.R.L., Campulung Muscel
  - Colentina Clinical Hospital, Cluj-Napoca
  - Rehabilitation Clinical Hospital, Cluj-Napoca
  - Timisoara Emergency County Clinical Hospital, Timișoara
- Russia (3):
  - Republican Clinical Hospital for Rehabilitation Treatment, Kazan'
  - Research Medical Complex Vashe Zdorovie, Kazan'
  - City Clinical Hospital 4, Saransk
- Serbia (5):
  - Clinical Center of Serbia, Belgrade
  - Clinical Hospital Centar Zvezdara, Belgrade
  - Military Medical Academy, Belgrade
  - Clinical Hospital Centre Zemun, Belgrade
  - Clinical Center Kragujevac, Kragujevac
- Spain (2):
  - Hospital Donostia, Donostia / San Sebastian
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- Ukraine (7):
  - Municipal Medical & Preventive Institution Chernigiv Regional Clinical Hospital, Chernihiv
  - Municipal Institution Dnipropetrovsk Regional Clinical Hospital na I.I. Mechnykov, Dnipropetrovsk
  - Regional Clinical Hospital, Ivano-Frankivsk
  - State Treatment and Prevention Institution Central Clinical Hospital of Ukrzaliznytsya, Kharkiv
  - Municipal Institution of Kyiv Regional Council Kyiv Regional Clinical Hospital, Kyiv
  - Volyn Regional Clinical Hospital, Lutsk
  - Municipal Institution Vinnytsya Regional Psychoneurological Hospital na OI Yushchenko, Vinnytsia

REFERENCES:
- [Result] Cohen JA, Arnold DL, Comi G, Bar-Or A, Gujrathi S, Hartung JP, Cravets M, Olson A, Frohna PA, Selmaj KW; RADIANCE Study Group. Safety and efficacy of the selective sphingosine 1-phosphate receptor modulator ozanimod in relapsing multiple sclerosis (RADIANCE): a randomised, placebo-controlled, phase 2 trial. Lancet Neurol. 2016 Apr;15(4):373-81. doi: 10.1016/S1474-4422(16)00018-1. Epub 2016 Feb 12. PMID 26879276
- [Result] Cohen JA, Comi G, Arnold DL, Bar-Or A, Selmaj KW, Steinman L, Havrdova EK, Cree BA, Montalban X, Hartung HP, Huang V, Frohna P, Skolnick BE, Kappos L; RADIANCE Trial Investigators. Efficacy and safety of ozanimod in multiple sclerosis: Dose-blinded extension of a randomized phase II study. Mult Scler. 2019 Aug;25(9):1255-1262. doi: 10.1177/1352458518789884. Epub 2018 Jul 25. PMID 30043658

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 55 study centers in 13 countries including the United States, Europe and Russia. Participants with multiple sclerosis (MS) were recruited between September 2012 and October 2013.
  The study consisted of a 24-week placebo-controlled treatment period and an optional 96-week blinded extension period.
Pre-assignment Details: Participants were randomly assigned in a 1:1:1 ratio to receive one of two daily doses of ozanimod (0.5 mg or 1 mg) or matching placebo for 24 weeks. Those who completed 24 weeks could enter a blinded extension phase and continue on their assigned doses of ozanimod, whereas those assigned to placebo were re-randomized in a 1:1 ratio to ozanimod 0.5 mg or 1 mg. In both periods the randomization was stratified by country.
Groups:
- Placebo: Participants received placebo capsules by mouth (PO) daily during the 24-week placebo-controlled treatment period.
- Ozanimod 0.5 mg: Participants received ozanimod 0.5 mg capsules PO daily during the 24-week placebo-controlled treatment period. Participants were given the option to enter into a blinded extension phase and continued to receive ozanimod 0.5 mg capsules PO daily for an additional 96 weeks of treatment.
- Ozanimod 1 mg: Participants received ozanimod 1 mg capsules PO daily during the 24-week placebo-controlled treatment period. Participants were given the option to enter into a blinded extension phase and continued to receive ozanimod 1 mg capsules PO daily for an additional 96 weeks of treatment.
- Placebo / Ozanimod 0.5 mg: Participants initially randomized to placebo during the 24-week placebo controlled treatment period were re-randomized to receive ozanimod 0.5 mg PO daily during the blinded extension period for 96 weeks.
- Placebo / Ozanimod 1 mg: Participants initially randomized to placebo during the 24-week placebo controlled treatment period were re-randomized to receive ozanimod 1 mg PO daily during the blinded extension period for 96 weeks.
Period: Placebo-controlled Treatment Period
Arm/Group | Placebo | Ozanimod 0.5 mg | Ozanimod 1 mg | Placebo / Ozanimod 0.5 mg | Placebo / Ozanimod 1 mg
Started | 88 | 87 | 83 | 0 | 0
Completed | 85 | 85 | 82 | 0 | 0
Not Completed | 3 | 2 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 1 | 0 | 0
Period: Blinded Active Extension Period
Arm/Group | Placebo | Ozanimod 0.5 mg | Ozanimod 1 mg | Placebo / Ozanimod 0.5 mg | Placebo / Ozanimod 1 mg
Started (Three participants who completed the placebo-controlled treatment period declined to enter the blinded extension period.) | 0 | 85 | 81 | 41 | 42
Completed | 0 | 75 | 75 | 37 | 36
Not Completed | 0 | 10 | 6 | 4 | 6
Not completed — Adverse Event | 0 | 1 | 0 | 2 | 2
Not completed — Lack of Efficacy | 0 | 0 | 2 | 0 | 2
Not completed — Physician Decision | 0 | 3 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 2 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 6 | 2 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population is defined as all randomized participants who received at least 1 dose of study drug; participants were analyzed according to the treatment they were randomized to receive and not according to what they actually received, if different.
Groups:
- Ozanimod 0.5 mg: Participants received ozanimod 0.5 mg capsules PO daily during the 24-week placebo-controlled treatment period.
- Ozanimod 1 mg: Participants received ozanimod 1 mg capsules PO daily during the 24-week placebo-controlled treatment period.
- Total: Total of all reporting groups
Arm/Group | Placebo | Ozanimod 0.5 mg | Ozanimod 1 mg | Total
Number analyzed (Participants) | 88 | 87 | 83 | 258
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.0 (8.67) | 38.1 (9.17) | 38.4 (9.82) | 38.5 (9.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 60 | 59 | 181
  Male | 26 | 27 | 24 | 77
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 87 | 84 | 83 | 254
  Black | 1 | 2 | 0 | 3
  Asian | 0 | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  North America | 4 | 4 | 4 | 12
  Western Europe | 6 | 4 | 3 | 13
  Eastern Europe | 78 | 79 | 76 | 233
Country of Enrollment [Count of Participants; unit: Participants]
  Poland | 44 | 44 | 44 | 132
  Serbia | 12 | 12 | 13 | 37
  Ukraine | 9 | 10 | 9 | 28
  Russia | 6 | 7 | 6 | 19
  United States | 4 | 4 | 4 | 12
  Romania | 2 | 2 | 2 | 6
  Georgia | 2 | 2 | 1 | 5
  Bulgaria | 2 | 1 | 1 | 4
  Greece | 1 | 1 | 2 | 4
  Spain | 2 | 1 | 1 | 4
  Italy | 2 | 1 | 0 | 3
  Belgium | 1 | 1 | 0 | 2
  Hungary | 1 | 1 | 0 | 2
Age at Multiple Sclerosis Diagnosis [Mean (Standard Deviation); unit: years] | 33.9 (8.30) | 34.8 (10.01) | 34.4 (9.51) | 34.4 (9.27)
Time Since Multiple Sclerosis Diagnosis [Mean (Standard Deviation); unit: years] | 4.6 (5.12) | 2.8 (4.98) | 3.6 (4.43) | 3.7 (4.90)
Expanded Disability Status Scale (EDSS) Score at Baseline [Mean (Standard Deviation); unit: units on a scale] — The EDSS is a scale for quantifying disability in MS. Eight functional systems (visual, brain stem, pyramidal, cerebellar, sensory, bowel & bladder, cerebral, and other functions) are scored on a scale from 0 (no disability) to 5 or 6 (more severe disability). Ambulation is also scored. Based on scores in the 8 functional systems plus gait, an overall score ranging from 0 (normal) to 10 (death due to MS) in 0.5 unit increments is assigned. Participants with EDSS scores of 0.0 to 4.5 are fully ambulatory; patients with EDSS scores of 5.0 to 9.5 have impaired ambulation.
  units on a scale | 2.85 (1.273) | 2.94 (1.287) | 2.86 (1.213) | 2.88 (1.255)
Time Since MS Symptom Onset [Mean (Standard Deviation); unit: years] | 8.1 (6.97) | 6.0 (6.41) | 6.2 (5.79) | 6.8 (6.47)
Number of Relapses Within the Last 12 months Prior to Screening [Mean (Standard Deviation); unit: relapses] | 1.3 (0.64) | 1.5 (1.18) | 1.3 (0.73) | 1.4 (0.88)
Number of Relapses Within the Last 24 months Prior to Screening [Mean (Standard Deviation); unit: relapses] | 1.8 (1.01) | 2.0 (1.79) | 1.9 (1.05) | 1.9 (1.33)
Number of Gadolinium Enhancing (GdE) Lesions [Mean (Standard Deviation); unit: lesions] — A lesion appearing on magnetic resonance imagery (MRI), following injection of the chemical compound gadolinium, that reveals a breakdown in the blood-brain barrier. This breakdown of the blood-brain barrier indicates either a newly active lesion or the re-activation of an old one.
  lesions | 1.4 (3.36) | 0.9 (1.42) | 1.3 (2.75) | 1.2 (2.64)

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Gadolinium-Enhancing (GdE) Lesions Assessed on Brain Magnetic Resonance Imaging (MRI) From Week 12 to Week 24
Description: The cumulative number of total GdE lesions on MRI from Week 12 to Week 24. MRI scans were assessed and scored by an independent MRI analysis center with no knowledge of treatment assignment or outcomes.
Time Frame: From Week 12 to Week 24; MRI was performed at Weeks 12, 16, 20, and 24
Population: The ITT population is defined as all randomized participants who received at least 1 dose of study drug.
  Missing data were imputed using the last valid non-missing, post-baseline observation which was carried forward if the participant was only missing 1 or 2 consecutive post-baseline scans. If there were no post-baseline data or the participant was missing > 2 consecutive scans, the mean number of lesions from participants in the same treatment group and visit was used as the imputed value.
Measure: Mean (Standard Deviation); unit: lesions
Groups:
- Placebo: Participants received placebo capsules PO daily during the 24-week placebo-controlled period.
Arm/Group | Placebo | Ozanimod 0.5 mg | Ozanimod 1 mg
Number analyzed (Participants) | 88 | 87 | 83
lesions | 11.1 (29.87) | 1.9 (4.77) | 1.5 (3.44)
Statistical Analysis 1: Comparison: Placebo vs Ozanimod 1 mg; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney) — To account for multiple comparisons, each of the 2 treatment comparisons was tested at the alpha = 0.04944 level of significance to keep the overall level of significance at 0.05; Wilcoxon-Mann-Whitney test stratified by absence or presence of gadolinium-enhancing lesions at Baseline
Statistical Analysis 2: Comparison: Placebo vs Ozanimod 0.5 mg; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]; Wilcoxon-Mann-Whitney test stratified by absence or presence of gadolinium-enhancing lesions at Baseline

2. Secondary Outcome: The Number of Gadolinium-Enhancing Lesions on Brain MRI Scan at Week 24
Description: MRI scans were assessed and scored by an independent MRI analysis center with no knowledge of treatment assignment or outcomes.
Time Frame: Week 24
Population: The ITT population is defined as all randomized participants who received at least 1 dose of study drug. Missing GdE data values were imputed using the mean number of lesions from participants in the same treatment group at the same visit.
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Placebo | Ozanimod 0.5 mg | Ozanimod 1 mg
Number analyzed (Participants) | 88 | 87 | 83
lesions | 3.2 (9.81) | 0.4 (1.27) | 0.2 (0.59)
Statistical Analysis 1: Comparison: Placebo vs Ozanimod 1 mg; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney); Wilcoxon-Mann-Whitney test stratified by absence or presence of gadolinium-enhancing lesions at Baseline
Statistical Analysis 2: Comparison: Placebo vs Ozanimod 0.5 mg; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney); Wilcoxon-Mann-Whitney test stratified by absence or presence of gadolinium-enhancing lesions at Baseline

3. Secondary Outcome: The Total Number of New or Enlarging Hyperintense T2-Weighted Brain MRI Lesions From Week 12 to Week 24
Description: The cumulative number of new or enlarging hyperintense T2-weighted brain MRI lesions from Week 12 to Week 24.
  MRI scans were assessed and scored by an independent MRI analysis center with no knowledge of treatment assignment or outcomes.
Time Frame: Week 12 to Week 24; MRI was performed at Weeks 12, 16, 20, and 24
Population: The ITT population is defined as all randomized participants who received at least 1 dose of study drug. Missing new or enlarging T2 data values were imputed using the mean from participants of the same treatment group at the same visit.
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Placebo | Ozanimod 0.5 mg | Ozanimod 1 mg
Number analyzed (Participants) | 88 | 87 | 83
lesions | 9.0 (20.87) | 1.4 (3.21) | 0.8 (1.86)
Statistical Analysis 1: Comparison: Placebo vs Ozanimod 1 mg; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney); Wilcoxon-Mann-Whitney test stratified by absence or presence of gadolinium-enhancing lesions at Baseline
Statistical Analysis 2: Comparison: Placebo vs Ozanimod 0.5 mg; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney); Wilcoxon-Mann-Whitney test stratified by absence or presence of gadolinium-enhancing lesions at Baseline

4. Secondary Outcome: Adjusted Annualized Relapse Rate (ARR) at Week 24
Description: A relapse was defined as new or worsening neurological symptoms attributable to MS and preceded by a relatively stable or improving neurological state for at least 30 days. Symptoms must have persisted for > 24 hours and not be attributable to confounding clinical factors. Relapses were confirmed when accompanied by objective neurological worsening based on examination by the blinded evaluator, consistent with an increase of ≥ 0.5 on the overall EDSS score relative to the most recent EDSS assessment, or 2 points on one of the functional system scale scores, or 1 point on ≥ two functional system scale scores.
  Relapse rate was calculated as the total number of confirmed relapses divided by the total number of days in the study * 365.
  ARR was based on a Poisson regression model, adjusted for region, relapses within 24 months before the study, and presence of gadolinium-enhancing lesions at Baseline.
Time Frame: Week 24
Population: The ITT population is defined as all randomized participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: relapses/year
Arm/Group | Placebo | Ozanimod 0.5 mg | Ozanimod 1 mg
Number analyzed (Participants) | 88 | 87 | 83
relapses/year | 0.50 [0.22 to 1.15] | 0.35 [0.15 to 0.82] | 0.24 [0.09 to 0.61]
Statistical Analysis 1: Comparison: Placebo vs Ozanimod 1 mg; Test type: Superiority; p = 0.0531, Poisson regression model; Adjusted for region, the number of relapses within 24 months prior to the study, and the absence or presence of GdE lesions at Baseline; Rate Ratio = 0.47, 95% CI 2-sided [0.22 to 1.01] — Rate ratio = Ozanimod / Placebo
Statistical Analysis 2: Comparison: Placebo vs Ozanimod 0.5 mg; Test type: Superiority; p = 0.2714, Poisson regression model; [statistical method as in outcome 4, analysis 1]; Rate Ratio = 0.69, 95% CI 2-sided [0.36 to 1.34] — Rate ratio = Ozanimod / Placebo

5. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAE) During the Placebo-Controlled Treatment Period
Description: An adverse event (AE) is any untoward medical occurrence that does not necessarily have a causal relationship with the investigational product (IP), including an abnormal laboratory finding, symptom or disease temporally associated with the use of an IP whether or not considered related to the IP. Serious AEs were events that resulted in death, were life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability or incapacity, were congenital abnormalities/birth defects, or important medical events which may have required medical intervention to prevent one of the above outcomes.
  The investigator assessed the severity of AEs as mild, moderate, or severe, and the relationship of each AE to treatment as unrelated, unlikely, possible, probable, or related based on timing and other known factors such as clinical state, environment, or other therapies.
Time Frame: From first dose of study drug up to Week 24, or up to 28 days after the last dose for participants who did not enter the extension period.
Population: Safety population was defined as all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ozanimod 0.5 mg | Ozanimod 1 mg
Number analyzed (Participants) | 88 | 87 | 83
Participants
  Any TEAE | 52 | 57 | 47
  Any moderate or severe TEAE | 23 | 23 | 13
  Any severe TEAE | 1 | 2 | 1
  Any TEAE related to study drug | 1 | 1 | 0
  Any serious TEAE | 0 | 3 | 0
  Any serious TEAE related to study drug | 0 | 0 | 0
  Any TEAE leading to discontinuation of study drug | 0 | 0 | 0
  Any death related to study drug | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAE) During Ozanimod Exposure
Description: AEs are reported from the start of the placebo-controlled period for participants originally assigned to ozanimod and from the start of the extension period for participants who switched to ozanimod after Week 24.
  Serious AEs were events that resulted in death, were life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability or incapacity, were congenital abnormalities/birth defects, or important medical events which may have required medical intervention to prevent one of the above outcomes.
  The investigator assessed the severity of AEs as mild, moderate, or severe, and the relationship of each AE to treatment based on timing and other known factors such as clinical state, environment, or other therapies.
Time Frame: From the first dose of ozanimod, either in the placebo-controlled or the blinded extension period, up to 4 weeks after the last dose; mean duration of exposure was 25.4, 30.9, 24.6, and 32.3 months in each treatment group respectively.
Population: Safety population was defined as all participants who received at least one dose of study drug in the blinded extension phase
Measure: Count of Participants; unit: Participants
Groups:
- Placebo / Ozanimod 0.5 mg: Participants initially randomized to placebo during the 24-week placebo controlled treatment period were re-randomized to receive ozanimod 0.5 mg capsules PO daily during the blinded extension period for 96 weeks.
- Ozanimod 0.5 mg: Participants received ozanimod 0.5 mg capsules PO daily during the 24-week placebo-controlled treatment period. Participants were given the option to enter into a blinded extension period and continued to receive ozanimod 0.5 mg capsules PO daily for an additional 96 weeks.
- Placebo / Ozanimod 1 mg: Participants initially randomized to placebo during the 24-week placebo controlled treatment period were re-randomized to receive ozanimod 1 mg capsules PO daily during the blinded extension period for 96 weeks.
- Ozanimod 1 mg: Participants received ozanimod 1 mg capsules PO daily during the 24-week placebo-controlled treatment period. Participants were given the option to enter into a blinded extension period and continued to receive ozanimod 1 mg capsules PO daily for an additional 96 weeks.
Arm/Group | Placebo / Ozanimod 0.5 mg | Ozanimod 0.5 mg | Placebo / Ozanimod 1 mg | Ozanimod 1 mg
Number analyzed (Participants) | 41 | 85 | 42 | 81
Participants
  Any TEAE | 26 | 73 | 32 | 61
  Any moderate or severe TEAE | 17 | 42 | 18 | 35
  Any severe TEAE | 2 | 4 | 1 | 2
  Any TEAE related to study drug | 2 | 3 | 1 | 3
  Any serious TEAE | 2 | 10 | 3 | 6
  Any serious TEAE related to study drug | 0 | 0 | 0 | 0
  Any TEAE leading to discontinuation of study drug | 2 | 1 | 1 | 0
  Any death related to study drug | 0 | 0 | 0 | 0

7. Post Hoc Outcome: Number of Gadolinium-Enhancing (GdE) Lesions During the Extension Period
Description: as for outcome 2
Time Frame: Weeks 24, 48, 72, and 120
Population: Participants who entered the blinded extension period, received at least 1 dose of study drug, and had any post-baseline assessment in the blinded extension period. Includes participants with non-missing MRI results at each time point.
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Placebo / Ozanimod 0.5 mg | Ozanimod 0.5 mg | Placebo / Ozanimod 1 mg | Ozanimod 1 mg
Number analyzed (Participants) | 41 | 85 | 42 | 81
lesions
  Week 24 (start of extension period) | 4.5 (13.02) | 0.4 (1.28) | 1.9 (5.93) | 0.2 (0.60)
  Week 48: number analyzed (Participants) | 38 | 80 | 40 | 79
  Week 48 | 0.6 (2.63) | 0.4 (1.30) | 0.4 (1.35) | 0.2 (0.56)
  Week 72: number analyzed (Participants) | 38 | 76 | 37 | 79
  Week 72 | 0.4 (1.95) | 0.4 (1.41) | 0.1 (0.28) | 0.2 (0.56)
  Week 120: number analyzed (Participants) | 37 | 72 | 36 | 74
  Week 120 | 0.1 (0.46) | 0.4 (1.49) | 0.1 (0.37) | 0.2 (0.51)

8. Post Hoc Outcome: Total Number of New or Enlarging Hyperintense T2-Weighted Brain MRI Lesions In the Extension Period
Description: The cumulative number of new or enlarging hyperintense T2-weighted brain MRI lesions from Week 12 to Week 24 in the placebo controlled period (reference) and during the first and second years of the extension period.
  MRI scans were assessed and scored by an independent MRI analysis center with no knowledge of treatment assignment or outcomes.
Time Frame: Weeks 12 to 24 of the placebo-controlled period and Week 24 to 72 (first year) and Week 72 - 120 (second year) in the extension period
Population: Participants who entered the blinded extension period, received at least 1 dose of study drug, and had any post-baseline assessment in the blinded extension period. Includes participants with non-missing MRI results in each time period.
Measure: Mean (Standard Error); unit: lesions
Arm/Group | Placebo / Ozanimod 0.5 mg | Ozanimod 0.5 mg | Placebo / Ozanimod 1 mg | Ozanimod 1 mg
Number analyzed (Participants) | 41 | 85 | 42 | 81
lesions
  Week 12 to 24 | 10.8 (3.58) | 1.4 (0.35) | 7.3 (3.07) | 0.9 (0.21)
  Week 24 to 72: number analyzed (Participants) | 38 | 76 | 37 | 79
  Week 24 to 72 | 4.3 (1.99) | 2.8 (0.72) | 1.5 (0.39) | 1.9 (0.84)
  Week 72 to 120: number analyzed (Participants) | 37 | 71 | 36 | 74
  Week 72 to 120 | 3.2 (1.31) | 2.3 (0.61) | 1.9 (0.48) | 0.7 (0.16)

ADVERSE EVENTS:
Time Frame: Placebo-controlled period: From first dose of study drug up to Week 24, or up to 28 days after the last dose for participants who did not enter the extension period. Extension period: From the first dose of ozanimod in the blinded extension period, up to 4 weeks after the last dose; up to 96 weeks.
Groups:
- Placebo-Controlled Period: Placebo: Participants received placebo capsules PO daily during the 24-week placebo-controlled period.
- Placebo-Controlled Period: Ozanimod 0.5 mg: Participants received ozanimod 0.5 mg capsules PO daily during the 24-week placebo-controlled period.
- Placebo-Controlled Period: Ozanimod 1.0 mg: Participants received ozanimod 1 mg capsules PO daily during the 24-week placebo-controlled period.
- Extension Period: Ozanimod 0.5 mg: Participants received ozanimod 0.5 mg capsules PO daily during the blinded extension period (Weeks 25 to 120).
- Extension Period: Ozanimod 1.0 mg: Participants received ozanimod 1 mg capsules PO daily during the blinded extension period (Weeks 25 to 120).
Arm/Group | Placebo-Controlled Period: Placebo | Placebo-Controlled Period: Ozanimod 0.5 mg | Placebo-Controlled Period: Ozanimod 1.0 mg | Extension Period: Ozanimod 0.5 mg | Extension Period: Ozanimod 1.0 mg
All-Cause Mortality (participants affected / at risk) | 0/88 | 0/87 | 0/83 | 0/126 | 0/123
Serious Adverse Events (participants affected / at risk) | 0/88 | 3/87 | 0/83 | 10/126 | 9/123
Other Adverse Events (participants affected / at risk) | 24/88 | 24/87 | 10/83 | 52/126 | 43/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo-Controlled Period: Placebo (N=88) | Placebo-Controlled Period: Ozanimod 0.5 mg (N=87) | Placebo-Controlled Period: Ozanimod 1.0 mg (N=83) | Extension Period: Ozanimod 0.5 mg (N=126) | Extension Period: Ozanimod 1.0 mg (N=123)
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Acute Myocardial Infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Irritable Bowel Syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Proctitis Infectious (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Clavicle Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Cauda Equina Syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Intracranial Aneurysm (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Optic Neuritis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Somatoform Disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Urethral Stenosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Menometrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Ovarian Cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Uterine Cervical Squamous Metaplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Uterine Haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Stasis Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo-Controlled Period: Placebo (N=88) | Placebo-Controlled Period: Ozanimod 0.5 mg (N=87) | Placebo-Controlled Period: Ozanimod 1.0 mg (N=83) | Extension Period: Ozanimod 0.5 mg (N=126) | Extension Period: Ozanimod 1.0 mg (N=123)
Nasopharyngitis (Infections and infestations) | 12 | 11 | 5 | 17 | 17
Upper Respiratory Tract Infection (Infections and infestations) | 3 | 4 | 3 | 20 | 11
Urinary Tract Infection (Infections and infestations) | 2 | 6 | 2 | 7 | 4
Alanine Aminotransferase Increased (Investigations) | 0 | 3 | 4 | 10 | 12
Gamma-Glutamyltransferase Increased (Investigations) | 0 | 2 | 5 | 11 | 8
Back Pain (Musculoskeletal and connective tissue disorders) | 9 | 5 | 2 | 5 | 7
Headache (Nervous system disorders) | 8 | 5 | 3 | 7 | 9
Hypertension (Vascular disorders) | 1 | 1 | 2 | 8 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator shall have the right to publish and/or present study data provided that the investigator shall (i) furnish the sponsor a copy of any proposed publication or presentation generally thirty (30) days in advance of the submission, (ii) delete any confidential information of the sponsor, and (iii) delay submission for generally up to ninety (90) days to permit the preparation and filing of intellectual property applications or until sponsor gives its consent in a timely manner.

DOCUMENTS (2):
  • Statistical Analysis Plan (2014-05-20): https://cdn.clinicaltrials.gov/large-docs/93/NCT01628393/SAP_000.pdf
  • Study Protocol (2014-10-01): https://cdn.clinicaltrials.gov/large-docs/93/NCT01628393/Prot_001.pdf